CLINICAL TRIAL: NCT00947388
Title: A Phase I Trial of Bendamustine Plus Alemtuzumab for the Treatment of Fludarabine Refractory Chronic Lymphocytic Leukemia
Brief Title: Bendamustine Plus Alemtuzumab for Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No more eligible patients
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1907; NCI-2010-00272 (Other: NCI/CTRP)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma
Keywords: Refractory Chronic Lymphocytic Leukemia; Bendamustine; Alemtuzumab; Phase I; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine plus Alemtuzumab (Experimental)
  Interventions: Drug: Bendamustine Hydrochloride; Biological: Alemtuzumab

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Bendamustine 70 mg/m2 IV Day 8 and 9 every 28 days for 6 courses of therapy
  Other Names: cytostasan hydrochloride; Ribomustin; SDX-105; Treanda
Biological: Alemtuzumab — Given subcutaneously (SC)on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26.
  Other Names: anti-CD52 monoclonal antibody; Campath; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52

SUMMARY:
This phase I trial is studying the side effects and best dose of alemtuzumab when given together with bendamustine hydrochloride in treating patients with relapsed chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that did not respond to fludarabine phosphate. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as alemtuzumab, can also block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bendamustine hydrochloride together with alemtuzumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of the combination of alemtuzumab and bendamustine (bendamustine hydrochloride) in patients with advanced CLL.

II. Establish the maximum tolerated dose of alemtuzumab up to the standard dose of 30mg thrice weekly when combined with bendamustine at a standard dose of 70 mg/m^2 day 8 and 9 monthly.

III. Define a recommended dose for subsequent Phase II studies. IV. Evaluate preliminary evidence of activity as determined by response rates with correlation to EAS flow cytometry.

OUTLINE: This is a dose-escalation study of alemtuzumab.

Patients receive bendamustine hydrochloride intravenously (IV) over 30-60 minutes on days 8 and 9 for up to 6 courses in the absence of disease progression or unacceptable toxicity and alemtuzumab subcutaneously (SC) on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CLL or SLL as defined by the WHO classification system with indications for treatment by National Cancer Institute (NCI) Working Group criteria.
2. Measurable disease (lymphocytes equal or greater than 5,000/µL, or measurable lymphadenopathy, or bone marrow involvement greater than 30%).
3. Males and females 18 years of age or older.
4. Patients must be relapsed or refractory and have been treated with a minimum of one prior purine analog-based chemotherapy regimen (e.g., fludarabine, cladribine, or pentostatin).
5. All previous cancer therapies, radiation, hormonal therapy and surgery, must have been discontinued at least 28 days prior to the start of treatment. Any cytotoxic chemotherapy must have been discontinued 28 days prior to the start of treatment. Acute toxicities from prior therapy must have resolved to Grade ≤ 1 above baseline.
6. Normal oxygen saturation with pulse oximetry on room air.
7. Hemoglobin 9 or greater gm/dL (may be post-transfusion).
8. Platelet count 50 x103/mL or greater
9. Total bilirubin less than 2 X ULN, and ALT and AST less than 2 x ULN.
10. Serum creatinine 2 X ULN or less. In addition, the calculated glomerular filtration rate (GFR) must be > 30cc/min.
11. ECOG Performance Status 2 or less.
12. Anticipated survival of at least 3 months.
13. For men and women of child-producing potential, use of effective contraceptive methods during the study and for one month after discontinuation of treatment.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Severe chronic obstructive pulmonary disease with hypoxemia or an uncorrectable pulmonary compromise.
3. Seizures not controlled by anticonvulsant therapy.
4. Participation in any investigational drug study within 28 days before study entry.
5. Patients with second malignancy requiring active treatment.
6. Active, symptomatic bacterial, fungal, or viral infection including active HIV or viral (A, B, or C) hepatitis.
7. Clinically significant bleeding event within the last 3 months, unrelated to trauma, or underlying condition that would be expected to result in a bleeding diathesis.
8. Patients with life- or function-threatening CLL complications (e.g., cord compression, hemolytic crisis, urinary tract obstruction).
9. Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any of the study's endpoints.
10. Systemic treatment for CLL/SLL within 28 days of study entry
11. Subjects with a history of leukemic meningitis, or signs and symptoms suggestive of leukemic meningitis, must have a negative lumbar puncture within 2 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the combination of alemtuzumab and bendamustine in patients with advanced CLL | up to 1 year
  AEs will be graded according to the NCI CTCAE, Version 3.0.

SECONDARY OUTCOMES:
Establish the maximum tolerated dose of alemtuzumab up to the standard dose of 30mg thrice weekly when combined with bendamustine at a standard dose of 70 mg/m2 day 8 and 9 monthly. | up to 12 weeks
  Adverse events (AEs) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0.
Clinical activity and response of the combination of bendamustine hydrochloride and alemtuzumab | up to 1 year
  Examined by summarizing response overall and by cohort as frequency counts and percentages. Response criteria as described by the National Cancer Institute-sponsored Working Group Guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Kalaycio, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Paolo Caimi, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio